CLINICAL TRIAL: NCT01474551
Title: A Single Center Phase II Trial of Vemurafenib (R05185426) in Poor Performance Status Patients With Unresectable Locally Advanced or Metastatic Melanoma Harboring a V600E/K Mutation
Brief Title: Vemurafenib (R05185426) in Poor Performance Status Patients With Unresectable Locally Advanced or Metastatic Melanoma Harboring a V600E/K Mutation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-091
Record Dates: First submitted 2011-11-15; First posted 2011-11-18 (Estimated); Results first posted 2015-04-30 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-10

CONDITIONS: Melanoma
Keywords: Vemurafenib; skin cancer; Stage IV; advanced stage III; 11-091
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — Vemurafenib

ARMS (1):
- vemurafenib (Experimental): This is a single institution phase II trial in stage III or IV melanoma patients with poor ECOG performance status (3 or 4). Patients must have melanoma with a BRAFV600E or BRAFV600K or mutation with measurable disease not curable by surgery.
  Interventions: Drug: vemurafenib

INTERVENTIONS:
Drug: vemurafenib — All patients would be treated with vemurafenib given orally at 960 mg twice a day, which was the phase III dose. One cycle is 4 weeks long.

SUMMARY:
The purpose of this study is to find out what effects, good and/or bad, vemurafenib has on the patient and the melanoma. Specifically, the investigators want to know how well vemurafenib shrinks melanoma. The investigators also want to find out how well vemurafenib can improve how well the patient functions.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old.
* Histologic proof of melanoma reviewed and confirmed by MSKCC.
* A confirmed EBRAFV600E or KBRAFV600K mutation.
* Stage IV melanoma, or advanced stage III not curable by surgery. Patients with active CNS metastases will be allowed on the study.
* Measurable disease by RECIST v1.1.
* ECOG performance status 3 or 4. The basis for the grading of performance is strict; there must be clear justification of the performance status grade (e.g. patient is confined to bed > 50% of time, or cannot carry out ADLs, or is otherwise disabled by burden of disease such as requiring supplemental O2).
* Patients must be able to swallow pills
* Adequate hematologic, hepatic and renal function as defined by the following:
* Absolute Neutrophil Count ≥ 1.0 x 109/L
* Hemoglobin ≥8.0g/dL, occasional transfusions are acceptable as vemurafenib does not have significant hematologic toxicities.
* Total bilirubin ≤2.0x the upper limit of normal, ≤3.0x the upper limit of normal if the patient has Gilbert's Syndrome.
* Alkaline phosphatase ≤2.0x the upper limit of normal.
* AST and ALT ≤2.0x the upper limit of normal.
* Serum creatinine ≤ 1.5x the upper limit of normal.

Exclusion Criteria:

* Uveal melanoma as primary.
* Concurrent chemotherapy, immunotherapy, or radiotherapy.
* Prior treatment with a RAF inhibitor. Other prior chemotherapy, immunotherapy, or radiotherapy will be allowed including prior treatment with a MEK inhibitor Patients must have had complete recovery from any adverse events or toxicities of prior cancer-directed therapies.
* Pregnant or lactating women.
* A second active malignancy. Prior malignancy will be allowed as long as the patient is known to be free of disease for at least 2 years. Patients with indolent B-cell malignancies will not be eligible.
* QTc interval > 500 msec.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Chapman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Alloo A, Garibyan L, LeBoeuf N, Lin G, Werchniak A, Hodi FS Jr, Flaherty KT, Lawrence DP, Lin JY. Photodynamic therapy for multiple eruptive keratoacanthomas associated with vemurafenib treatment for metastatic melanoma. Arch Dermatol. 2012 Mar;148(3):363-6. doi: 10.1001/archdermatol.2011.3080. PMID 22431777
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual: 11/15/2011 Protocol Closed to Accrual: 03/12/2013 Primary Completion Date (if applicable): 03/12/2013 Recruitment Location is the medical clinic
Period: Overall Study
Arm/Group | Vemurafenib
Started | 2
Completed | 1
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Vemurafenib
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Objective Response
Description: The Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 will be used to determine treatment response. In order to be considered evaluable for response, a patient must have completed at least 1 cycle of therapy. Patients who do not complete a cycle of therapy can be replaced.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Vemurafenib
Number analyzed (Participants) | 1
participants
  Stable Disease | 1
  Complete Response | 0
  Partial Response | 0
  Progression of Disease | 0

ADVERSE EVENTS:
Arm/Group | Vemurafenib
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vemurafenib (N=2)
Creatinine increase (Investigations) | 1 (1)
Death NOS (General disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vemurafenib (N=2)
Blood bilirubin increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (8)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (14)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (6)
INR increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes